CLINICAL TRIAL: NCT04228627
Title: Intravenous Iron for Non-anaemic Iron Deficiency in Pregnancy:a Multicenter,Two-arm,Randomised Controlled Trial
Brief Title: Ferritin Screening And IRon Treatment for Maternal Anemia and FGR Prevention Trial
Acronym: FAIR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Collaborators: Allama Iqbal Medical College (Other); Universidad de Granada (Other); Fatima Jinnah Medical University (Other)
Responsible Party: Principal Investigator, Tayyiba Wasim, Professor, Services Institute of Medical Sciences, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB/2019/599/SIMS
Record Dates: First submitted 2020-01-09; First posted 2020-01-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Iron Deficiency (Without Anemia); Pregnancy Related
Keywords: anemia, ferritin
MeSH Terms: conditions — Iron Deficiencies; Anemia

STUDY DESIGN:
Intervention Model Description: Multi centre randomised trial
Who Masked: Investigator
Masking Description: Allocation concealment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Active Comparator): Intravenous Iron to correct Iron deficiency without anaemia
  Interventions: Drug: Parentral Iron
- Prophylaxis (No Intervention): Usual antenatal care

INTERVENTIONS:
Drug: Parentral Iron — Correction of Iron stores without anaemia
  Arms: Treatment

SUMMARY:
Prevalence of anemia in Asia is more than 50%. All woman who book for antenatal care with non-anaemic iron deficiency (NAID) can be offered therapeutic doses of parentral iron, as a directly observed complete therapy, to prevent of maternal anaemia and fetal growth restriction. The investigators will compare this intervention with usual care in a multicentre randomised trial.

DETAILED DESCRIPTION:
Prevalence of anemia (haemoglobin less than 11 gm/dl) in Asia is more than 50% and non-anaemic iron deficiency (ferritin less than 30 microgm/l) or NAID is likely to be more prevalent than this figure. It has been hypothesised that NAID in pregnancy can be linked to maternal fatigue and anaemia, and infant birth weight and growth restriction. The investigators will compare, in NAID, active intervention (therapeutic doses of parentral iron, as a directly observed complete therapy, to replenish iron stores) vs usual care (prophylactic oral iron supplementation) to prevent of maternal anaemia and fetal growth restriction in a multicentre randomised trial.

ELIGIBILITY:
Inclusion Criteria:

* Non-anaemic iron deficiency

Exclusion Criteria:

* Anaemia or normal iron stores

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Maternal anaemia | 36 weeks' gestation
  Haemoglobin concentration (g/dl)

SECONDARY OUTCOMES:
Fetal growth restriction | At birth
  Birthweight for gestational age (percentile)

CONTACTS AND LOCATIONS:
Overall Officials: TAYYIBA Wasim, Principal Investigator — Services Institute of Medical Sciences, Pakistan
Locations (3):
- Pakistan (3):
  - Fatima Jinnah Medical University, Lahore, Punjab Province
  - TAYYIBA Wasim, Lahore, Punjab Province
  - Allama Iqbal Medical College, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: Yes
On completion of study we will happily discuss data sharing with any legitimate party with an IPD meta-analysis protocol.
Supporting Information: Study Protocol
Time Frame: Following publication of study
Access Criteria: An acceptable IPD meta-analysis protocol with a suitable data sharing agreement

REFERENCES:
- [Background] Pratt JJ, Khan KS. Non-anaemic iron deficiency - a disease looking for recognition of diagnosis: a systematic review. Eur J Haematol. 2016 Jun;96(6):618-28. doi: 10.1111/ejh.12645. Epub 2015 Sep 17. PMID 26256281
- [Background] Wasim T, Bushra N, Tajammul A, Humayun S, Rasool S, Shahbaz F, Riaz A, Siddique F, Khawaja KI, Fatima A, Zafar Z, Khan KS. Ferritin screening and Iron treatment for maternal anemia and fetal growth restriction prevention - A multicenter randomized controlled trial (FAIR Study). Pak J Med Sci. 2023 Jan-Feb;39(1):293-299. doi: 10.12669/pjms.39.1.6686. PMID 36694741
- [Derived] Wasim T, Bushra N, Nasrin T, Humayun S, Tajammul A, Khawaja KI, Irshad S, Fatima S, Yasin A, Zamora J, Cano-Ibanez N, Fernandez-Felix BM, Khan KS; Ferritin screening and iron treatment for maternal anaemia and fetal growth restriction prevention (FAIR) Study Group. Intravenous iron for non-anaemic iron deficiency in pregnancy: a multicentre, two-arm, randomised controlled trial. Lancet Haematol. 2026 Jan;13(1):e22-e29. doi: 10.1016/S2352-3026(25)00315-1. PMID 41482443